CLINICAL TRIAL: NCT03409055
Title: Pleural Effusions Are Associated With Adverse Outcomes After Cardiac Surgery
Brief Title: Pleural Effusions After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, Prof. Dr. med. Dr. rer. nat., MSc, Charite University, Berlin, Germany
Other Study IDs: PONTOS-Effusions
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Pleura; Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 0: patients without pleural effusion
- Group 1: patients with pleural effusion
- Group 2: patients with pleural Effusion and need of drainage

SUMMARY:
Pleural effusions occur commonly in patients recovering from cardiac surgery, however, the impact on outcomes is not well characterized. The purpose of this study is to characterize the outcomes of cardiac surgery patients with pleural effusions.

All patients undergoing cardiac surgery between 2006 and 2019 were included in this observational, cross-sectional analysis using propensity matching.

DETAILED DESCRIPTION:
Pleural effusions are common in patients recovering from cardiac surgery. Symptomatic patients with pleural effusions complain of shortness of breath, cough, chest pain and are more hypoxic and tachypneic. Clinically significant effusions can slow recovery in the hospital and beyond, and are a critical source of hospital readmissions after discharge. It is not well characterized how this impacts hospital outcomes. Further it is unknown if the effusions themselves are associated with impaired outcomes, or if pleural effusions simply arise in more complicated, older patients, thus suggesting the impaired outcomes are the result of coexisting morbidities. To better understand the impact of this complication and to address the question mentioned before, this study was carried out to determine the clinical and economic outcomes of pleural effusions in propensity-matched patients during early recovery from cardiac surgery. To compare patient groups with and without pleural effusion, the following baseline characteristics were used: e.g. age, sex, body-mass-index, priority of surgery, type of surgery, duration of surgery, APACHE II Score of patients on admission in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* In-patients of the Charité Universitätsmedizin Berlin
* at least 18 years old
* female or male sex
* cardiosurgical intervention (OPS 5.35 and 5.36) between 01/06 and 12/19
* post-operative monitoring in the intensive care unit

Exclusion Criteria:

* previous cardiosurgical interventions during the same hospital stay
* incomplete documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male and female patients who have undergone cardiac surgery in the period 01/06-12/19 at Campus Mitte in the Charité, approx. 11,000 patients.
Sampling Method: Probability Sample
Enrollment: 11198 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | an average of 30 days
  In-Hospital mortality
hospital stay | an average of 30 days
  Length of hospital stay

SECONDARY OUTCOMES:
Need of drainage | an average of 30 days
  Incidence of drainage in patients with pleural effusions
extubation | an average of 15 hours
  time to extubation
renal replacement | an average of 30 days
  incidence of renal replacement therapy
transfusions | an average of 30 days
  number of transfusions needed
ICU stay | an average of 15 days
  Length of Intensive Care Unit (ICU) stay

CONTACTS AND LOCATIONS:
Overall Officials: Felix Balzer, MD, MSc, PhD, Principal Investigator — Charite Universitätsmedizin Berlin
Locations (1):
- Charité - Universitaetsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Schiefenhovel F, Poncette AS, Boyle EM, von Heymann C, Menk M, Vorderwulbecke G, Grubitzsch H, Treskatsch S, Balzer F. Pleural effusions are associated with adverse outcomes after cardiac surgery: a propensity-matched analysis. J Cardiothorac Surg. 2022 Dec 7;17(1):298. doi: 10.1186/s13019-022-02050-y. PMID 36476289